CLINICAL TRIAL: NCT00526565
Title: Randomized Trial of Tapas Acupressure for Weight Loss Maintenance
Acronym: LIFE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AT003928-01A1 (NIH); R01AT003928-01A1 (NIH)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TAT (Tapas Acupressure Technique)
  Interventions: Behavioral: Tapas Acupressure Technique
- 2 (Active Comparator): SS (Professionally facilitated social support groups)
  Interventions: Behavioral: Social support

INTERVENTIONS:
Behavioral: Tapas Acupressure Technique — Practice of the TAT technique involves application of pressure to select acupoints combined with specific mental focus. The TAT pose involves lightly touching the tips of the left thumb and 4th finger to the area 1/8 inch above the inner corner of each eye and the 3rd finger to the point midway between the eyes, about ½ inch above eyebrow level. The right hand is on the back of the head, with the palm cradling the occiput and the thumb just above the hairline. Once in this position, the process is to 1) focus attention on the identified problem or behavior to be changed (e.g., over-eating); 2) focus on a positive thought related to the problem; 3) focus on the thought of healing or clearing the origins of the problem; and 4) focus on an awareness of healing or clearing any storage of the problem, at a cellular, mental, emotional, or energetic level.
  Other Names: TAT
  Arms: 1
Behavioral: Social support — The LIFE SS maintenance intervention will consist of a series of professionally facilitated social support groups where the session content is directed by the participants. The contact hours for SS will match those of the TAT intervention. The initial SS group session will orient participants to the basics of weight maintenance, and subsequent sessions will provide opportunities for participants to share experiences and ask questions. Participants may choose to use behavioral tools as desired. In addition to the basic materials about weight loss maintenance used in both maintenance interventions, will we use the materials already used in the weight loss program for the SS group as needed. We will measure adherence by taking attendance at the SS group sessions.
  Other Names: Social support groups
  Arms: 2

SUMMARY:
This randomized clinical trial evaluates the efficacy of TAT(Tapas Acupressure Technique) compared to a Social Support (SS) group for the primary outcome of weight loss maintenance. We recruit obese adults from the Kaiser Permanente Northwest managed care setting. Those who meet eligibility criteria are entered into an intensive six-month weekly group-based behavioral weight loss program. Those who meet threshold weight loss criteria (n=~288) are randomly assigned to either TAT instruction or social support group. Participants in both groups attend the same schedule of group meetings with parallel contact hours. Participants in the TAT group are advised to practice the technique at home. Participants are weighed and questionnaires administered at entry, randomization, and at 12 and 18 months post entry. The main outcome measure is weight at 18 months.

ELIGIBILITY:
* Inclusion criteria for the Phase I weight loss program:

  * Men and women
  * At least 30 years of age
  * BMI 30-50 kg/m2 (inclusive)
  * Weight <400 lbs
  * Reside in Portland metropolitan area including Vancouver/Clark County, Washington
  * Willing and able to participate in all aspects of the intervention
  * Willing to attend the group-based weight loss program for 6 months
  * Willing to follow a reduced calorie healthy dietary pattern
  * Willing to exercise on a regular basis
  * Willing to lose 10 pounds during the 6-month weight loss program
  * Willing to accept random assignment to one of the two maintenance interventions
  * Willing to provide informed consent

Exclusion criteria for the Phase I weight loss program

* Medical conditions or treatments that would be contraindicated using a diet and exercise weight loss treatment
* Treatment for cancer (except for non-melanoma skin cancer) currently or in the past 2 years
* Diabetes treated with insulin; does not exclude diet-controlled, controlled with sulfonylurea (glyburide, glipizide, etc.) with primary physician's approval, or controlled with other oral agents (metformin, precose, glitazone.)
* Psychiatric hospitalization in past 2 years
* Conditions that require limitation of physical activity
* Congestive heart failure
* Cardiovascular disease (stroke, MI, CABG, angioplasty/stent) in the past 2 years
* Taking weight loss medications currently or within past 6 months
* Any history of weight loss surgery or scheduled surgery for weight loss.
* Liposuction in the past 12 months
* Prior acupuncture or acupressure treatments for weight loss
* Planning to leave the area prior to the end of the program
* Body weight change > 20 pounds in the past 6 months
* Pregnant, breast feeding, or planning pregnancy prior to the end of participation
* Current participation in another clinical trial
* Investigator discretion for safety or adherence reasons
* Household member (living at the same address) of another participant in this study
* LIFE clinical trial staff member or family member of LIFE trial staff person

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
weight | 18 months

SECONDARY OUTCOMES:
psychosocial measures, exercise, food frequency, and food cravings variables | randomization, and @ months 12 and 18

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Elder, MD, Principal Investigator — Kaiser Permanente

REFERENCES:
- [Derived] Elder CR, Gullion CM, Debar LL, Funk KL, Lindberg NM, Ritenbaugh C, Meltesen G, Gallison C, Stevens VJ. Randomized trial of Tapas Acupressure Technique for weight loss maintenance. BMC Complement Altern Med. 2012 Mar 15;12:19. doi: 10.1186/1472-6882-12-19. PMID 22417316